CLINICAL TRIAL: NCT03566498
Title: The Effect Of Immediate Versus Early Oral Hydration On Caesarean Section Post Operative Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Shafy El Shahawy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMOH
Record Dates: First submitted 2018-06-01; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate hydration (Experimental): They will be allowed to start oral fluids immediately (within the first 2 hours post operatively) beginning with water or clear fluids (but not milk or soda containing drinks), the amounts will be according to their needs, solid food will be given gradually after tolerating the drinks and intravenous fluids will be given beside all of that and till the return of intestinal movements.
  Interventions: Dietary Supplement: Immediate hydration
- Early hydration (Active Comparator): They will receive the routine intravenous fluids and the oral fluids will be given after 8 hours post operatively and gradually, solid food will be allowed after that gradually too and the intravenous fluids will be stopped after return of intestinal movements.
  Interventions: Dietary Supplement: Early hydration

INTERVENTIONS:
Dietary Supplement: Immediate hydration — They will be allowed to start oral fluids immediately (within the first 2 hours post operatively) beginning with water or clear fluids (but not milk or soda containing drinks), the amounts will be according to their needs, solid food will be given gradually after tolerating the drinks and intravenous fluids will be given beside all of that and till the return of intestinal movements
  Arms: Immediate hydration
Dietary Supplement: Early hydration — They will receive the routine intravenous fluids and the oral fluids will be given after 8 hours post operatively and gradually, solid food will be allowed after that gradually too and the intravenous fluids will be stopped after return of intestinal movements.
  Arms: Early hydration

SUMMARY:
The aim of this study is to evaluate the effect of immediate oral hydration initiated within 2 hours after uncomplicated Caesarean section

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of immediate oral hydration initiated within 2 hours after uncomplicated Caesarean section on the following post-operative outcomes:

1. Post-operative nausea, vomiting, abdominal distention and abdominal cramps.
2. Return of intestinal movements.
3. Duration of intravenous fluid administration.
4. Duration of hospital stay.
5. Participant satisfaction

ELIGIBILITY:
Inclusion Criteria:

* • Uncomplicated pregnancy.

  * Uncomplicated elective or emergency Caesarean section under regional anesthesia

Exclusion Criteria:

* • Having medical disorders in the form of: hypertension, DM, and Hepatic disorders.

  * Having bleeding disorders.
  * Having intraoperative bowel or bladder injury.
  * Having intraoperative or immediate postoperative severe bleeding.
  * Having chronic gastrointestinal problems, like chronic constipation, peptic ulcer, esophagitis, hiatus hernia or irritable bowel syndrome.
  * Having abdominal adhesions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Postpartum vomiting | 48 hours
  through a questionnaire patients were asked if they had vomiting or not and the nomber of attacks of vomitting

SECONDARY OUTCOMES:
Return of intestinal movements | 24 hours
  through physical examination and auscultation of the intestinal sounds
Duration of intravenous fluid administration | 24 hours
Duration of hospital stay | 48 hours
Participant satisfaction | 48 hours
  through a questionnaire patients were asked about degree of satisfaction
  1- satisfied 2- neutral 3- not satisfied